CLINICAL TRIAL: NCT03428503
Title: Comparison of Efficacy of Intravenous Paracetamol and Dexketoprofen for Acute Traumatic Musculoskeletal Pain in the Emergency Department: A Double-Blinded, Randomized, Controlled Trial
Brief Title: Comparison of Efficacy of Intravenous Paracetamol and Dexketoprofen for Acute Traumatic Musculoskeletal Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ibrahim Turkcuer, Professor, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015HZL031
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Musculoskeletal Pain
Keywords: paracetamol; dexketoprofen; emergency department; musculoskeletal pain
MeSH Terms: conditions — Musculoskeletal Pain; Emergencies | interventions — Acetaminophen; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Experimental): 1000 mg of paracetamol (perfalgan 10mg/ml solution Bristol-Myers Squibb_UK) intravenous (IV) was given 100 patients
  Interventions: Drug: Paracetamol
- Dexketoprofen (Experimental): Second group: dexketoprofen 50 MG (Arveles ampoule -Ufsa- Istanbul) intravenous (IV) was given 100 patients
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Paracetamol — 1000 mg of paracetamol (perfalgan 10mg/ml solutionBristol-Myers Squibb_UK) intravenous (IV) was given 100patients
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Dexketoprofen — Second group: dexketoprofen 50 MG (Arveles ampoule -Ufsa- Istanbul) intravenous (IV) was given 100 patients
  Other Names: ASEKET; DARKIN; DEXALGIN; DESTIYO; DEXCORIL
  Arms: Dexketoprofen

SUMMARY:
* Currently, paracetamol and nonsteroidal antiinflammatory drugs are widely used by emergency physicians in Turkey for the treatment of patients with acute traumatic musculoskeletal pain.
* The objective of the study is compare the efficacy of intravenous dexketoprofen with paracetamol in the treatment of acute traumatic musculoskeletal pain.

DETAILED DESCRIPTION:
* This is the randomized double blinded clinical trial to compare the efficacy of these two drugs in this clinical setting.
* A randomized clinical trial was conducted in the Emergency Department (ED) of Pamukkale University Medical Faculty Hospital
* Study personnel (emergency physicians and nurses) were trained before the study.
* When intravenous drugs (Paracetamol, Dexketoprofen) was being recommended, an eligibility checklist was completed by the attending physician.
* If there were no exclusion criteria, written informed consent was obtained and baseline information, including initial acute traumatic musculoskeletal pain severity ratings with visual analog scale (VAS) were recorded.
* The need for identification and enrollment of participants by staff with conflicting work pressures resulted in recruitment of a convenience sample of patients.
* All patients eligible for the study were randomized to one of two groups:

First Group: 1000 mg of paracetamol ( perfalgan 10mg/ml solutionBristol-Myers Squibb_UK) intravenous (IV) was given 100 patients, Second Group: dexketoprofen 50 mg ( arveles ampoule -Ufsa- Istanbul) intravenous (IV) was given 100 patients which determined to be applied as a group.

Drug packs prepared in 150 ml serum physiology were numbered by an independent nurse, who not involved in the study.

* Drugs were prepared according to the computer-generated random number sequence to assign treatment allocations
* The allocation list was kept by the emergency nurse. Patients received the paracetamol, dexketoprofen medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug pack was obtained, and administered intravenously.
* Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms)
* One researcher blinded to patient allocation observed the whole procedure and recorded the acute non-traumatic musculoskeletal pain scores.
* Patients in both groups received two types of medication in a similar manner, thus ensuring double blind.
* Acute traumatic musculoskeletal pain scores were recorded at 0, 15, 30 and 60 min on a VAS of 1 to 10
* Rescue medication (Fentanyl 1mcg/kg) was given intravenous to patients if pain VAS scores ≥ 5 in sixty minutes after study drug administration.
* All other medications required during the study also were recorded.
* During the study, pulse rate, systolic blood pressure, diastolic blood pressure, respiration rate and oxygen saturation (SpO2) were recorded at baseline (0 min), 15, 30, and 60 min.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were aged 18 years or older, 65 years or younger
* Isolated traumatic musculoskeletal pain
* Patients who agree to work and receive the approval
* VAS (visual analog scale) score>5.

Exclusion Criteria:

* Patients with severe liver, kidney,pulmonary and cardiac heartfailure
* To be Pregnancy and breast-feeding
* Have received analgesics in the last 6hours
* Patients of childbearing age who are not using a birth control method.
* Patients with neurological deficits
* Patients with sciatica and back pain
* Patients with cardiac chest pain
* Patients with chronic pain
* Patients with pre-existing dexketoprofen and paracetamol-induced gastrointestinal bleeding and perforation
* Patients with reflected pain
* Patients with neoplastic pain
* Patients with an allergy trait (paracetamol and dexketoprofen)
* Illiterates and patients with vision problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Decrement of the pain on VAS | Baseline and 60 minutes
  Comparison of the reduction of traumatic musculoskeletal pain VAS (visual analog scale) score between the two groups. - (First group Paracetamol and Second Dexketoprofen)

CONTACTS AND LOCATIONS:
Overall Officials: Atakan Yilmaz, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz A, Sabirli R, Ozen M, Turkcuer I, Erdur B, Arikan C, Demirozogul E, Sarohan A, Seyit M, Ok N. Intravenous paracetamol versus dexketoprofen in acute musculoskeletal trauma in the emergency department: A randomised clinical trial. Am J Emerg Med. 2019 May;37(5):902-908. doi: 10.1016/j.ajem.2018.08.023. Epub 2018 Aug 8. PMID 30100336